CLINICAL TRIAL: NCT06649929
Title: Nuestro Sueno: Cultural Adaptation of a Couples Intervention to Improve Positive Airway Pressure Adherence and Sleep Health Among Latino Couples With Implications for Alzheimer's Disease Risk
Brief Title: Nuestro Sueno: Cultural Adaptation of a Couples Intervention to Improve PAP Adherence and Sleep Health Among Latino Couples With Implications for Alzheimer's Disease Risk
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Arizona (Other); Banner Health (Other)
Responsible Party: Principal Investigator, Kelly Glazer Baron, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00177835; 4R33AG084477-02 (NIH)
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Sleep Apnea; Sleep Disturbance
Keywords: sleep; couples; positive airway pressure
MeSH Terms: conditions — Sleep Apnea Syndromes; Parasomnias

STUDY DESIGN:
Intervention Model Description: Couples will be randomized 1:1 to intervention and control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Couples-based treatment- Patient (Experimental): In this group, couples will attend 3-telehealth based sessions with a community health worker for education and interventions to improve communication, sleep quality and PAP use
  Interventions: Behavioral: Couples-based treatment- Patient
- Couples-based treatment- Partner (Experimental): In this group, couples will attend 3-telehealth based sessions with a community health worker for education and interventions to improve communication, sleep quality and PAP use
  Interventions: Behavioral: Couples-based treatment- Partner
- Information Control- Patient (Active Comparator): In this group, couples will recieve a standardized packet of insomnia about obstructive sleep apnea and starting positive airway pressure.
  Interventions: Other: Information control- Patient
- Information Control- Partner (Active Comparator): In this group, couples will recieve a standardized packet of insomnia about obstructive sleep apnea and starting positive airway pressure.
  Interventions: Other: Information control- Partner

INTERVENTIONS:
Behavioral: Couples-based treatment- Patient — couples will attend 3-telehealth based sessions to provide eduction, increase self-efficacy and teach skils based in principles of brief behavioral therapy for insomnia
  Arms: Couples-based treatment- Patient
Behavioral: Couples-based treatment- Partner — couples will attend 3-telehealth based sessions to provide eduction, increase self-efficacy and teach skils based in principles of brief behavioral therapy for insomnia
  Arms: Couples-based treatment- Partner
Other: Information control- Patient — Information only plus treatment as usual
  Arms: Information Control- Patient
Other: Information control- Partner — Information only plus treatment as usual
  Arms: Information Control- Partner

SUMMARY:
The goal of this clinical trial is to learn if the culturally adapted couples sleep health intervention (Nuestro Sueno) improves positive airway pressure use and sleep among Hispanic couples in which one partner was diagnosed with sleep apnea and starting positive airway pressure treatment.

The main questions are:

1. Does Nuestro sueno improve the patient's positive airway pressure use over the first 3 months of using it compared to an information control?
2. Does Nuestro sueno improve sleep quality for both the patient and partner, compared to an information control?
3. Does Nuestro sueno improve other aspects of life including quality of life and memory, compared to an information control?

DETAILED DESCRIPTION:
Latino adults in the United States are 1.5 times more likely to develop Alzheimer's disease and related dementias compared to non-Hispanic white adults. Obstructive sleep apnea affects 9.8% of Latino adults and confers a five-fold increased risk of Alzheimer's disease diagnosis. Consequences also extend to the bedpartner, as bedpartners of those with obstructive sleep apnea experience significant sleep disturbances, including sleep fragmentation and 3 times greater risk of insomnia. Given solid mechanistic links between both obstructive sleep apnea and insomnia and Alzheimer's Disease risk, effective obstructive sleep apnea treatment has the potential to promote healthy cognitive aging and reduce Alzheimer's Disease risk for both partners. While the front-line treatment for obstructive sleep apnea, positive airway pressure, is highly effective at reducing obstructive sleep apnea symptoms and may reduce or forestall Alzheimer's Disease risk, its potential is severely diminished, as up to 80% of patients are non-adherent. Extant positive airway pressure adherence interventions are limited in that they are exclusively focused on the individual, neglecting to consider the role of the bedpartner in treatment, and developed primarily in non-Hispanic white populations. Therefore, there is a critical need to develop evidence-based, and culturally-adapted interventions that address the impact of obstructive sleep apnea and its treatment on both partners and within a culturally-tailored framework. The goal of this study is to develop and test "Nuestro Sueño" a culturally-adapted intervention to promote positive airway pressure adherence and sleep health among Latino couples. This study will involve a randomized clinical trial to evaluate the feasibility, treatment satisfaction and preliminary efficacy of Nuestro Sueño versus information control in a sample of 80 patients with obstructive sleep apnea and their partners (i.e., 40 couples per treatment arm) across two sites (Utah and Arizona). The intervention focuses specifically on the interpersonal mechanisms of enhancing dyadic coping and communication, using intervention materials resonant with cultural beliefs and values. If successful, Nuestro Sueño, an innovative and culturally-adapted intervention, has the potential to significantly advance the treatment of obstructive sleep apnea, and may elucidate a critical, modifiable target of prevention and intervention to promote healthy aging and reduce disparities in Alzheimer's Disease risk among Latino couples.

ELIGIBILITY:
Patients inclusion criteria:

* Self-reported Latino ethnicity
* Age >35, 3)
* Diagnosed with obstructive sleep apnea and intend to start PAP
* Never used positive airway pressure or-restarting CPAP after 3 months
* Married or cohabiting with a romantic partner for >1 year
* Able to read/write English or Spanish
* Access to cellular (active data plan) or Wi-Fi, or able to use study devices in order to complete the telehealth intervention.

Partner inclusion criteria:

* Able to read/write in English or Spanish
* Interested in improving their sleep (yes/no)
* Access to cellular (active data plan) or Wi-Fi, to complete the telehealth intervention or able to use a study device.

Partners of all ethnicities will be invited to participate. The intervention will be delivered in couples preferred language.

Exclusion criteria for both patient and partner

* High risk or presence of moderate to severe comorbid sleep disorders (i.e., restless legs syndrome)
* History of cognitive or neurological or major psychiatric disorders
* Unstable or serious medical illness that would interfere with participation (cancer, renal disease on dialysis, moderate to severe chronic obstructive pulmonary disease
* Patients with need for more complex care (e.g., adaptive servo-ventilation, supplemental oxygen) or concurrent sleep apnea treatment such as bariatric surgery or oral appliance
* Overnight work > 1x per month; 7) Pregnancy/desire to become pregnant in the study period; 8) Current participation in behavioral sleep treatment (e.g., cognitive behavioral therapy for insomnia)
* Concurrent participation in another clinical trial
* Caregiving for an infant < 2 years old or adult who requires overnight assistance

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | 36 months
  Defined as the ability to achieve the recruitment goals of the study, to recruit approximately 3-4 couples per month over the study period

SECONDARY OUTCOMES:
Proportion of Days With positive airway pressure Use of 4 Hours or More | 3 months
  The primary efficacy measure for this pilot trial was the proportion of days that patients used CPAP for 4 hours or more over the first 3 months. This 4 hour cutoff was selected becasue it is the minimum usage defined by Medicare and other insurance companies. We obtained patients' CPAP usage by downloading data from their machine using a remote dashboard. Data are only available for patients because partners were not using the treatment. This variable is defined as a proportion, calculated as the number of days with CPAP usage of 4 hours or more divided by the total number of days collected in the 3 month recording period. Scores can range from 0 (no days with use to 1, indicating all days with use of 4 hours or more).
Self-reported Sleep Disturbance | 3 months
  Patient sleep quality on the Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance scale, 8 item, version 8b. Models evaluated change from baseline to 3 months. Raw are converted to t-scores, with a range of 28.9-76.5, a mean of 50 and a SD of 10. Higher scores indicate poorer sleep subjective quality.

OTHER OUTCOMES:
Intervention Completion | 1 month
  Percentage of participants who completed the intervention sessions: 3 sessions for the couples-based treatment group and 1 handout and phone call for the information control group
Retention | 3 months
  We defined retention as the number of participants completing the 3 month follow-up. Our goal was to acheive at least 85% retention.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Banner Health, Tucson, Arizona
  - University of Utah, Salt Lake City, Utah